CLINICAL TRIAL: NCT04261088
Title: Assisted Suicide in Switzerland
Status: Active, not recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999920059; 20-CC-N059
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12-02

CONDITIONS: Assisted Suicide
Keywords: Ethics; Switzerland; End of life; Assisted Death; Natural History
MeSH Terms: conditions — Suicide, Assisted; Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experts in Swiss assisted suicide: Persons in Switzerland who are experts in how assisted suicide is practiced. We will beexamining already collected interviews.

SUMMARY:
Background:

Researchers want to learn more about how the Swiss model of assisted suicide works. To do this, they have interviewed 25 Swiss experts. The researchers will draw on research in the fields of ethics, law, and medicine to analyze the transcripts.

Objective:

To describe the practice of assisted suicide in Switzerland and to study how the policy is carried out, how the right-to-die societies work, and the ethical implications of the practice.

Eligibility:

Swiss experts in the field of assisted suicide

Design:

The study includes 25 interviews that have already been conducted. The participants were:

* academics
* doctors and others in medical care
* a government official
* representatives of right-to-die societies.

Researchers will analyze the data using qualitative methods. Two researchers will develop a coding scheme and code the texts and analyze the data.

DETAILED DESCRIPTION:
Switzerland is the only country in the world that enables assisted suicide by lay people, i.e.,

people who are not physicians. All other countries that have adopted aid-in-dying legislation

require that a physician provides this assistance. This project probes the reasons for adopting this policy, and the advantages and the disadvantages of the Swiss model at the end of life. Are the Swiss aid-in-dying volunteers able to provide well-informed assistance to patients in need? Is the Swiss model one to be followed by other nations? The project will focus on the work of the Swiss aid-in-dying societies. The study draws on research in the fields of ethics, law and medicine. Its novelty lies in incorporating different methods of analysis, reflecting on the right to die with dignity within a liberal framework that aims to respect fundamental human rights.

ELIGIBILITY:
* INCLUSION/EXCLUSION:

The study includes 25 interviews with Swiss experts that have been conducted.

* Gender: Men 14, Women 11
* Backgrounds of interviewees: Academics 14, Physicians and other medical care 6, Right to die associations 4, Government official 1
* Race and ethnicity: All white Swiss.
* Age range: Unknown, but all are adults.
* No vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 transcripts of interviews with: Academics 14, Physicians and other medical care 6, Right to die associations 4, Government official 1
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive study | Ongoing
  This is a qualitative descriptive study of transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Y Kim, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States